CLINICAL TRIAL: NCT01392079
Title: A Prospective, Multi-center Phase II Study of Subcutaneous Alemtuzumab Combined With Oral Dexamethasone, Followed by Alemtuzumab Maintenance or Allogeneic Stem-cell Transplantation, in Chronic Lymphocytic Leukemia Which is Associated With 17p Deletion or is Refractory to Fludarabine
Brief Title: Subcutaneous Alemtuzumab Combined With Oral Dexamethasone, Followed by Alemtuzumab Maintenance or Allo-SCT in CLL With 17p- or Refractory to Fludarabine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: Technical University of Munich (Other); WiSP Wissenschaftlicher Service Pharma GmbH (Other); German CLL Study Group (Other)
Responsible Party: Principal Investigator, Stephan Stilgenbauer, Prof. Dr. med., University of Ulm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cll2O; 2007-003099-20 (EudraCT Number)
Record Dates: First submitted 2011-06-28; First posted 2011-07-12 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL; 17p deletion; refractory to fludarabine; subcutaneous alemtuzumab; CLL with 17p- or refractory to fludarabine
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Chromosome 17 deletion | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alemtuzumab (Experimental): 30 mg alemtuzumab will be administered subcutaneously 3 times weekly for 4 weeks (total of 12 doses of 30 mg alemtuzumab) with premedication (as needed) and infection prophylaxis; combined with oral dexamethasone 40 mg total dose for 4 days every 2 weeks; evaluation at end of cycle (i.e. after 12 doses of 30 mg alemtuzumab).
  If CR is documented after week 4 (12 doses of 30 mg alemtuzumab) or 8 (24 doses of 30 mg alemtuzumab), maintenance treatment with alemtuzumab or withdrawal from the study and stem cell transplantation will be instituted at this time point.
  After a maximum of three 4-week cycles (total of 36 doses of 30 mg alemtuzumab, in case of interruptions this may take longer than 12 weeks), maintenance treatment with alemtuzumab or withdrawal from the study and stem cell transplantation will be instituted. Maintenance treatment with alemtuzumab will continue for a maximum of two years, with evaluation every three months, unless there is PD.
  Interventions: Drug: Alemtuzumab

INTERVENTIONS:
Drug: Alemtuzumab — Alemtuzumab 30 mg s.c. 3 × weekly for 28 days (Days 1, 3, 5; 8, 10, 12; etc.)

SUMMARY:
Aims and objectives

* Assessment of the efficacy of the study treatment in the study population in terms of response rate, progression-free survival, failure-free survival and overall survival.
* Acquisition of further data to expand the data base on the toxicity of the study treatment.
* Assessment of the efficacy of the study treatment in biological risk groups.
* Assessment of response in terms of minimal residual disease. Number of patients and estimated duration Total no. of patients: 122 (~29 with 17p deletion for first-line therapy, ~29 with 17p deletion for second- or higher-line treatment, ~65 fludarabine-refractory irrespective of 17p status).

Duration for each patient: Max. 12 weeks of treatment in three 4-week cycles, then up to two years maintenance treatment.

DETAILED DESCRIPTION:
CLL refractory to therapy based on fludarabine or with 17p deletion has a poor prognosis. Patients with F-refractory CLL have a remission rate of 20% after various salvage regimens and a median overall survival (OS) of <12 months (Keating et al., 2002a). CLL patients with 17p deletion have a median OS of 16 months after first-line treatment with fludarabine or FC in the CLL4 trial of the GCLLSG (Figure 2; Stilgenbauer et al., 2005b; Eichhorst et al., 2006).

Alemtuzumab is the most active single agent in fludarabine-refractory CLL, with remission rates of 30-40% and median OS of 16-28 months (Keating et al., 2002b, Rai et al., 2002). Furthermore, alemtuzumab is of proven efficacy in CLL with 17p deletion and the subcutaneous administration is as effective as the intravenous application (Stilgenbauer & Döhner, 2002, Lozanski et al., 2004, Stilgenbauer et al., 2004).

However, the outcome of fludarabine-refractory CLL is still poor, owing to the facts that the majority of patients do not achieve a remission and that the average duration of remission is short. Therefore, the current trial aims at achieving: (i) a higher remission rate, by adding high-dose dexamethasone to alemtuzumab, and (ii) prolongation of remission duration and survival by alemtuzumab maintenance or allogeneic stem-cell transplantation (SCT). High-dose steroids have shown activity independently of 17p and p53 status, and are effective in debulking large lymph nodes, a weakness of alemtuzumab (Bellosillo et al., 2002, Thornton et al., 2003, Pettitt et al., 2006). Maintenance treatment with alemtuzumab improved remission duration in the CLL4B trial and allogeneic SCT resulted in disease control in high-risk CLL in the CLL3X trial (Wendtner et al., 2004, Dreger et al., 2005).

This is a prospective, open, multi-center Phase II study conducted by the Deutsche CLL Studiengruppe (DCLLSG; German CLL Study Group, GCLLSG). There will be only one treatment group and thus no randomization. The study will be conducted at approximately 40 investigation sites in Germany, Austria and France.

The study will be conducted according to the EG Directive on Good Clinical Practice, the German Arzneimittelgesetz (AMG, 12. Novelle) as well as - with respect to the local activities and regulations - to the corresponding laws in France and Austria.

A total of 122 patients (adults, males and females, in-patients and out-patients; 2 to 10 patients are expected to be recruited by each of the centers) will be recruited, with stratification by detailed diagnosis. The distribution of female and male patients is not relevant for the study as both sexes are affected by CLL and treatment effects are not different in both groups (GCP-V § 7, 2). Recruiting will stop when the 122th. patient has completed the first four-week cycle of treatment. The study will be concluded when the last patient has completed treatment with alemtuzumab according to this protocol. The retrieval of additional follow-up data may be appropriate to achieve mature data in the survival endpoints.

Subcutaneous alemtuzumab (30 mg) will be administered three times weekly (days 1, 3 and 5) along with oral dexamethasone (40 mg/day, days 1-4, every 2 weeks) for at least 4 weeks (corresponding to 12 doses of alemtuzumab, in case of treatment interruption this may take longer than 4 weeks) and, for patients who show at least SD, a maximum of 12 weeks (36 doses of alemtuzumab, in case of treatment interruption this may take longer than 12 weeks). Thereafter, maintenance therapy with alemtuzumab will be instituted for a maximum of two years. If CR (including bone marrow histology and imaging (chest X-ray and ultrasound, CT if indicated) is documented before week 12, i.e. after week 4 (12 doses of 30 mg alemtuzumab) or 8 (24 doses of 30 mg alemtuzumab), maintenance treatment with alemtuzumab will be instituted at this time point.

In this study it is recommended to start the dose of alemtuzumab directly at 30 mg. However, the dose of alemtuzumab can be increased gradually (3 mg day -2, 10 mg day -1 and 30 mg day 1, as in earlier studies), according to the investigators discretion.

Staging will be performed at inclusion to the study and after 12 doses of alemtuzumab (aim: at the end of Week 4), after 24 doses of alemtuzumab (aim: at the end of Week 8), and after 36 doses of alemtuzumab (aim: at the end of Week 12) of treatment. Patients showing progressive disease (PD) (according to NCI criteria) will be withdrawn from the study. If hematological or other toxicity is seen, treatment will be interrupted and the dose will be reduced according to the prescription information.

If after 12 weeks there is stable disease (SD), partial response (PR) or complete response (CR), then maintenance treatment will be given, with continued subcutaneous alemtuzumab (30 mg every 14 days). Patients for whom stem-cell transplantation is a realistic treatment option will be offered the possibility of receiving allogeneic stem-cell treatment in another clinical trial (CLLX2 or other GCLLSG trial). The latter will however only be offered if (1) the patient is eligible according to protocol and (2) a HLA-compatible donor is available who has given his/her informed consent. There should be a treatment-free period of at least 2 months before SCT, details are specified in the corresponding protocol.

Appropriate premedication and infection prophylaxis will be administered. After each disease staging (i.e. every three months during the maintenance phase), if there is SD, PR or CR, then patients will continue study therapy (alemtuzumab maintenance). Maintenance therapy will be stopped after two years.

During the study, continual monitoring of efficacy and toxicity will be performed. Early stopping rules will be applied if major intolerability is observed.

Response will be assessed by clinical examination, blood counts, clinical chemistry, chest X-ray (plain radiograph of the chest), ultrasound of the abdomen, CT scanning (if indicated), bone marrow cytology and histology (only in cases of possible CR), and assessment of MRD (for molecular response rate only). Time points for response evaluation according to NCI criteria will be after 12 doses, 24 doses, and 36 doses of alemtuzumab. For an uninterrupted treatment course, this will be after 4, 8 and 12 weeks respectively. (If treatment with alemtuzumab is interrupted, then the time points for all subsequent doses, assessments and other procedures will be delayed correspondingly; i.e., the number of doses is the determining factor for elapsed treatment time, and not the calendar date; see above, "Staging will be performed...".) Follow-up assessment will continue at three-month intervals for at least three years.

The following time schedule is anticipated for the study:

* Start of recruitment: January 2008
* End of recruitment: September 2011
* End of study procedures (conclusion of maintenance therapy): December 2013 (plus eventual additional follow-up)

ELIGIBILITY:
Inclusion Criteria:

1. The patient has CLL requiring treatment (Binet C or A/B with "active disease" according to the NCI criteria).
2. One or both of the following is true:

   * The patient's disease is refractory to a previous fludarabine-containing regimen, defined as no CR or PR according to NCI criteria, or progression within 6 months after a fludarabine-containing regime. (N.B.: Within the framework of this trial, the term "fludarabine-refractory" is synonymous to a refractory status to any established purine analogue (i.e. pentostatin, cladribine); this also encompasses bendamustine, as this drug molecule contains both an alkylating and a purine analogue moiety. Acc. to experimental findings and clinical experience, its mechanism of action differs distinctly from that of a pure alkylator (Cheson et al., 2009, Leoni et al., 2008)).
   * 17p deletion is present (irrespective of whether previously treated or untreated).
3. The patient is at least 18 years of age.
4. The patient's performance status is 0, 1 or 2 on the WHO/ECOG scale.
5. Any previous chemotherapy and/or immunotherapy ended at least four weeks before the first study treatment with alemtuzumab.
6. The patient has recovered from all previous chemotherapy and/or immunotherapy.
7. For fertile men and for women of childbearing potential: Adequate contraception (oral contraceptives, intrauterine device or barrier method in conjunction with spermicidal jelly).
8. The patient has given written informed consent to participate in the study.

Exclusion Criteria:

1. The patient has received more than five different prior therapeutic regimens.
2. Any major organ dysfunction is present (e.g. unstable angina pectoris, NYHA III/IV heart insufficiency, significant coronary stenoses, uncontrolled diabetes mellitus, uncontrolled hypertension, pulmonary disease with hypoxemia, renal failure).
3. Any of the following laboratory values are found at the screening visit to be >2 × the upper limit of the normal range: serum creatinine, serum bilirubin, ASAT, ALAT.
4. Any active infection is present.
5. B-PLL or Richter transformation is diagnosed or suspected (e.g. symptoms or cytology).
6. There is involvement of the central nervous system.
7. The patient is known to be positive for human immunodeficiency virus (HIV).
8. CMV viremia is present, as demonstrated by pp65 EA or CMV-DNA.
9. The patient has previously been treated with alemtuzumab. (Exception: alemtuzumab used in a "non-therapeutic" context, i.e. administered as part of a conditioning regimen prior to SCT).
10. The patient has received autologous or allogeneic SCT within the past six months.
11. The patient is receiving long-term systemic treatment with corticosteroids or has received such treatment in the four weeks before first treatment with alemtuzumab.
12. Any additional active malignancy is present.
13. The patient has ever had an anaphylactic response to humanized antibodies.
14. For female patients: The patient is pregnant or lactating.
15. The patient has a history of drug or alcohol abuse that might lead to inability to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2008-02; Primary Completion 2012-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Response rate | 2.5 years
  Time points for response evaluation according to NCI criteria will be:
  * The end of each treatment cycle: after 12 doses (4 weeks actual treatment), 24 doses (8 weeks actual treatment), and 36 doses (12 weeks actual treatment) of alemtuzumab
  * During maintenance therapy, every three months
  * During follow-up, every three months
  * A final response assessment will be made at the end of study treatment if the patient's participation is ended at a point other than one of those specified above.

SECONDARY OUTCOMES:
Progression-free-survival | up to five years
  Progression-free survival: time from study entry to the detection of progressive disease according to NCI criteria or death of any cause, whichever occurs first.
Failure-free survival | up to five years
  Failure-free survival: time from study entry until next treatment, detection of progressive disease according to NCI criteria or death of any cause, whichever occurs first.
Overall survival | up to five years
  Time from study entry to death of any cause.
Number of participants with Adverse Events as a measure of safety and tolerability | up to 2.5 years
  Acquisition of further data to expand the data base on the toxicity of the study treatment. (Type, frequency, severity, timing and relatedness of AEs and laboratory abnormalities observed during different treatment cycles)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Stilgenbauer, Prof Dr med, Principal Investigator — University of Ulm
Locations (38):
- Austria (2):
  - Hanuschkrankenhaus Wien, Vienna
  - University Hospital, Vienna
- France (15):
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Hopital Avicenne, Bobigny
  - CHU Estaing, Clermont-Ferrand
  - Hôpital Henri Mondor, Creteil -APHP, Créteil
  - CHU de Grenoble, Grenoble
  - CHU Claude Huriez, Lille
  - Hôpital Edouard Herriot Lyon, Lyon
  - CHU de Nancy, Nancy
  - CHU Nantes, Nantes
  - Hôpital Pitié Salpêtrière Paris-APHP, Paris
  - Hôpital Saint-Louis Paris -APHP, Paris
  - Centre Hospitalier Marechal Joffre Hôpital Saint-Jean Perpignan, Perpignan
  - CHU de Poitiers, Poitiers
  - CHU Robert-Debre, Reims
  - CHU de Tours, Tours
- Germany (21):
  - Charité CBF Berlin, Berlin
  - University of Cologne, Cologne
  - Dresden Universtiy Hospital, Dresden
  - Essen University, Essen
  - Freiburg University, Freiburg im Breisgau
  - Goettingen University, Göttingen
  - LMU Munich, Großhadern
  - AK St. Georg Hamburg, Hamburg
  - Hannover medical school (MHH), Hanover
  - Heidelberg University, Heidelberg
  - Homburg/Saar University, Homburg/Saar
  - Dr. Soeling Kassel, Kassel
  - Kiel University, Kiel
  - Mainz University, Mainz
  - TU Munich, Munich
  - Nuernberg University Hospital, Nuremberg
  - OncoProGbR Regensburg, Regensburg
  - Universtiy of Tuebingen, Tübingen
  - University of ulm, Ulm
  - Dr. Schlag Wuerzburg, Würzburg
  - University Hospital Wuerzburg, Würzburg

REFERENCES:
- [Derived] Edelmann J, Holzmann K, Tausch E, Saunderson EA, Jebaraj BMC, Steinbrecher D, Dolnik A, Blatte TJ, Landau DA, Saub J, Estenfelder S, Ibach S, Cymbalista F, Leblond V, Delmer A, Bahlo J, Robrecht S, Fischer K, Goede V, Bullinger L, Wu CJ, Mertens D, Ficz G, Gribben JG, Hallek M, Dohner H, Stilgenbauer S. Genomic alterations in high-risk chronic lymphocytic leukemia frequently affect cell cycle key regulators and NOTCH1-regulated transcription. Haematologica. 2020 May;105(5):1379-1390. doi: 10.3324/haematol.2019.217307. Epub 2019 Aug 29. PMID 31467127
- [Derived] Steinbrecher D, Jebaraj BMC, Schneider C, Edelmann J, Cymbalista F, Leblond V, Delmer A, Ibach S, Tausch E, Scheffold A, Bloehdorn J, Hallek M, Dreger P, Dohner H, Stilgenbauer S. Telomere length in poor-risk chronic lymphocytic leukemia: associations with disease characteristics and outcome. Leuk Lymphoma. 2018 Jul;59(7):1614-1623. doi: 10.1080/10428194.2017.1390236. Epub 2017 Oct 24. PMID 29063805